CLINICAL TRIAL: NCT03615937
Title: KeySteps@JC - Early Child Intervention for Underprivileged Families in Hong Kong
Brief Title: KeySteps@JC - Early Child Intervention
Acronym: KSJC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KeySteps@JC
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Lower Socioeconomic Background
MeSH Terms: interventions — Mass Screening; Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Intervention (Experimental): This is a holistic package of interventions, including:
  1. Child interactive intervention (dialogic reading and play intervention)
  2. Family Empowerment (positive parenting and grandparenting)
  3. Access to Community Hub and its services
  4. Enhancement to the kindergartens
  5. Health education, screening, and support
  Interventions: Behavioral: Child interactive intervention; Behavioral: Family Empowerment; Behavioral: Access to Community Hub and its services; Other: Enhancement to the kindergartens; Other: Health education, screening, and support
- Health Support (Active Comparator): This is a control arm with only health components.
  1. Health education, screening, and support
  Interventions: Other: Health education, screening, and support

INTERVENTIONS:
Behavioral: Child interactive intervention — The Child Interactive Intervention will be delivered through a Dialogic Reading Program, which is an individual/group level intervention component for both families and kindergartens. The original Dialogic Reading Program aims to enhance children's literacy and oral language skills by using the specific technique of shared book reading developed by Whitehurst and colleagues (1988). However, this project will expand from the original Dialogic Reading Program template to include alignment with local kindergarten curriculum and themed interactive activities that help build social competence and emotional maturity in children, in addition to cognitive skills.
  Arms: Comprehensive Intervention
Behavioral: Family Empowerment — Family empowerment in this project can be conceptualized across three main pillars: 1) adaptive parenting; 2) adaptive extended family environment; and 3) familial resources. Typically, adaptive parenting is translated into positive parenting programs for primary caregivers, and the rest of the family environment involves extended caregivers. However, families from disadvantaged environments encounter many hurdles that hinder effective parenting and relationship nurturing, and parents' mental wellbeing are also consistently impacted by competing demands.
  Arms: Comprehensive Intervention
Behavioral: Access to Community Hub and its services — A new model of Community Hub will be implemented and there will be two hubs established in two respective districts. The Community Hubs act as an alternative venue to implement service delivery of intervention packages, such as activity sessions in the Child Interactive Intervention, Parenting Program, and mentor-mentee experience exchange, which provide families institutional flexibility and extended support while internalizing new practices. There will also be health education, consultation support and developmental assessments. The Hubs will play the roles of promoting and interweaving play-based learning into the lives of families frequently faced with competing demands and a lack of resources, and enable a protracted network for parents.
  Arms: Comprehensive Intervention
Other: Enhancement to the kindergartens — This intervention package aims at providing a better physical and social kindergarten environment to maximize developmental reach and expedite timely interception and feedback without adding burden to teachers and frontline service professionals.
  Arms: Comprehensive Intervention
Other: Health education, screening, and support — Health seminars and interactive workshop will be provided to the families. Screen for common child health problems (e.g. dental and visual) will also be conducted. A support hotline and website will be established for the participants.

SUMMARY:
The proposed early intervention is grounded within a framework that incorporates two key aspects: a multi-level component with nested or layered contexts, and a growth aspect with early and on-going social investments to mitigate disparate trajectories among underprivileged children. Capital is built across multiple levels over a three-year period during the critical window of early childhood - among the young children themselves plus their primary caregivers and teachers (Level 1), the family unit and school environment (Level 2), and the larger community (Level 3) that includes infrastructure for extended learning and bridges with other resource institutions. Schools will be stratified and then randomized to receive an integrated multi-disciplinary intervention or a health consultation control. Evaluation will include a comprehensive battery to assess baseline capacity in children, parents, teachers, relationship characteristics between them, as well as the early learning environment at home and at school (Year 1), repeated measures to index intermediate (ongoing for specific individual and family domains, 3 months for school changes, annual progress reports) and final response (Year 3) to treatment, and age- and time-appropriate (e.g. age 4, 5, 6; stage of parenting; experience of teachers) indices of functioning at each annual checkpoint.

DETAILED DESCRIPTION:
Socioeconomic disadvantage permeates multiple levels of environmental contexts in which children are raised, including the family environment and schools. Disparities in life outcomes can be observed in early childhood and developmental gaps widen over time. Continued exposure to adverse conditions propagates the developing child on an increasingly risky trajectory. This study aims to mitigate the adverse effect of socioeconomic disadvantage on children and their families.

This is a clustered randomised controlled study recruiting 32 kindergartens in two underprivileged districts (16 in each district) in Hong Kong. District is a blocking factor. Within each district, 8 kindergartens will be randomised in comprehensive intervention group while the remaining 8 will be in health support group. The families in the comprehensive intervention will receive a holistic package of interventions, including child interactive intervention, family empowerment, and health support. The families in the health support group will only receive health support intervention.

In addition, a stepped wedge cluster randomised control trial design will be used to deliver and evaluate the health intervention package (health seminars/workshops, dental check-up/treatment, visual check-up/treatment). The schematic diagram of the design is shown in the figure below.

Another randomisation will be conducted to determine the sequence in which the health intervention takes place. 4 KGs will be provided with the health intervention in each month sequentially from Nov 2018 to Jun 2019 (totally 8 months). The randomisation should ideally be stratified by district (SSP/TSW) and the original group allocation (Comprehensive/Health). In other words, in each month, 1 KG from SSP Comprehensive, 1 from SSP Health, 1 from TSW Comprehensive, 1 from TSW Health will receive the health intervention package.

In analysis, the time exposed to intervention (e.g. Gp1 exposed to 8 months at Jun 2018) will be used to evaluate the effect of the intervention. Since the time exposed to intervention (i.e. the starting time of the intervention) is randomised, internal validity should be ensured. In addition, the stratification of district and the original group allocation should eliminate the influence of these factors.

ELIGIBILITY:
Inclusion Criteria:

1. K1 children [~3 years], with a selected Pre-Nursery group [~2 years], and their families attending participating kindergartens.
2. Kindergartens located at Sham Shui Po and Tin Shui Wai districts in Hong Kong based on the following criteria:

   1. Full-day program
   2. Pre-Primary Education Voucher Scheme
   3. Basic school facilities (minimally >1 classroom and a basic activity room available)
   4. Average school tuition fee in the past 5 years (<HKD 40,000)
   5. Proportion of teachers with early childhood education bachelor degrees or above. Teachers of participating children will be their facilitators/assessors in this study.

Exclusion Criteria:

1. Children and families from non-participating kindergartens; children below and above K1 (except for a selected Pre-Nursery group).
2. Non-English/Chinese speaking subjects.
3. Teachers of non-participating children and kindergartens.
4. Non-consenting subjects.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1216 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Child development | Three years after start of intervention
  Full scale score of Hong Kong Early Child Development Scale (HKECDS); The HKECDS includes items from the following eight subscales: Personal, Social and Self-Care (7 items), Language Development (13 items), Pre-academic Learning (27 items), Cognitive Development (10 items), Gross Motor (12 items), Fine Motor (9 items), Physical Fitness, Health and Safety (7 items), and Self and Society (10 items). The items are scored on a 0/1 basis. The subscale items can be summed to a total score. Higher score indicate better developmental outcomes.

SECONDARY OUTCOMES:
Physical health and well-being | Three years after start of intervention
  Aggregated score based on physical and health assessments such as body height and weight, blood pressure, spirometry, ultrasound measured bone density, and skin prick test using principal component analysis
Socio-emotional development | Three years after start of intervention
  Aggregated score based on validated tools such as Strength and Difficulties Questionnaires and Chinese Early Development Instrument using principal component analysis
Neurocognitive development | Three years after start of intervention
  Aggregated score based on validated tools such as Hong Kong Early Child Development Scale and Parents' Evaluation of Developmental Status using principal component analysis
Parental Capacity and Parenting Practices | Three years after start of intervention
  Aggregated score based on validated tools such as Parent-child Conflict Tactics Scale using principal component analysis
Parenting and developmental literacy | Three years after start of intervention
  Aggregated score based on validated tools such as Parent-Child Interaction Scale, Parenting Styles and Dimensions Questionnaire using principal component analysis
Parental mental health and emotion processing | Three years after start of intervention
  Aggregated score based on validated tools, such as General Self-Efficacy Scale, Connor Davidson Resilience Scale using principal component analysis
School readiness | Three years after start of intervention
  Total scale score of the Chinese Early Development Instrument using principal component analysis

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ip, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung C, Hui ANN, Wong RS, Rao N, Karnilowicz W, Chung K, Chan J, Ip P. Effectiveness of a Multicomponent Parenting Intervention for Promoting Social-Emotional School Readiness Among Children From Low-Income Families in Hong Kong: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2022 Apr 1;176(4):357-364. doi: 10.1001/jamapediatrics.2021.6308. PMID 35129606